CLINICAL TRIAL: NCT07278960
Title: Enhancing Algorithms for the Management of Children Conceived by Assisted Reproductive Technologies Based on a Comprehensive Assessment of the Impact of Modern Methods of Conception on Their Health Status
Brief Title: Enhancing Management Algorithms for Children Conceived Via Assisted Reproductive Technologies
Status: Recruiting | Type: Observational
Sponsor: Kazakhstan's Medical University "KSPH" (Other)
Collaborators: International Clinical Center for Reproductology "PERSONA" (Unknown)
Responsible Party: Principal Investigator, Sevara Ilmuratova, Senior researcher, Kazakhstan's Medical University "KSPH"
Other Study IDs: AP26100341
Record Dates: First submitted 2025-11-14; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Children; ART; Anthropometric Characteristics; Somatic Health Status; Neurological Condition; Urogenital Pathology
Keywords: ART; health status; children after ART; offspring; urogenital pathology; anthropometric charachteristics; neurological conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children born after ICSI: Anthropometric data: will include weight, height, and head and chest circumference at the time of examination. Birth anthropometric data will be sourced retrospectively, while the WHO Child Growth Standards will be utilized to evaluate weight, height, head, and chest circumference relative to age and gender.
  Psychomotor development: This evaluation will employ standardized instruments such as the R. Griffiths Mental Development Scale and Denver Developmental Screening Tests.
  Reproductive Health: The study will also evaluate the effect of ICSI, particularly in cases of male infertility, on the reproductive health and development of 200 male children under three years of age, in comparison with children conceived via classic IVF. This evaluation will involve objective examinations conducted by a pediatric andrologist to investigate the prevalence of urogenital pathology, , supplemented by ultrasounds of the scrotum, kidneys, and bladder.
  Interventions: Diagnostic Test: Inhibin B; Diagnostic Test: Anti-Müllerian Hormone (AMH)
- children born after IVF: Anthropometric data: will include weight, height, and head and chest circumference at the time of examination. Birth anthropometric data will be sourced retrospectively, while the WHO Child Growth Standards will be utilized to evaluate weight, height, head, and chest circumference relative to age and gender.
  Psychomotor development: This evaluation will employ standardized instruments such as the R. Griffiths Mental Development Scale and Denver Developmental Screening Tests.
  Reproductive Health: The study will also evaluate the effect of ICSI, particularly in cases of male infertility, on the reproductive health and development of 200 male children under three years of age, in comparison with children conceived via classic IVF. This evaluation will involve objective examinations conducted by a pediatric andrologist to investigate the prevalence of urogenital pathology, , supplemented by ultrasounds of the scrotum, kidneys, and bladder.
  Interventions: Diagnostic Test: Inhibin B; Diagnostic Test: Anti-Müllerian Hormone (AMH)

INTERVENTIONS:
Diagnostic Test: Inhibin B — The study will also evaluate the effect of ICSI, particularly in cases of male infertility, on the reproductive health and development of 200 male children under three years of age, in comparison with children conceived via classic IVF. This evaluation will involve objective examinations conducted by a pediatric andrologist to investigate the prevalence of urogenital pathology, supplemented by ultrasounds of the scrotum, kidneys, and bladder. Additionally, hormonal status will be assessed by Inhibin B and Anti-Müllerian Hormone (AMH). Anamnestic data will be collected to explore the relationship between the reproductive health of fathers and their sons born after ICSI.
Diagnostic Test: Anti-Müllerian Hormone (AMH) — The study will also evaluate the effect of ICSI, particularly in cases of male infertility, on the reproductive health and development of 200 male children under three years of age, in comparison with children conceived via classic IVF. This evaluation will involve objective examinations conducted by a pediatric andrologist to investigate the prevalence of urogenital pathology, supplemented by ultrasounds of the scrotum, kidneys, and bladder. Additionally, hormonal status will be assessed by Inhibin B and Anti-Müllerian Hormone (AMH). Anamnestic data will be collected to explore the relationship between the reproductive health of fathers and their sons born after ICSI.

SUMMARY:
Research Methods and Ethical Issues

1. Main Scientific Questions and Hypotheses of the Project The primary objective of this project is to investigate the impact of advanced ART methods on the health status of children. The central scientific questions being addressed include: What are the consequences of ICSI and FET on the physical, cognitive, and reproductive health of children? The underlying hypothesis posits that children conceived by advanced ART methods may present with health indicators that deviate from the established norms.
2. Description of the Experiments

Research Methods:

To achieve the goals of the study, the following stages are anticipated:

1. Retrospective Analysis of Anamnestic Data:

   This stage involves studying the relationship between the physical status and morbidity structure of 300 children under the age of three, who were conceived by advanced ART methods. Additionally, the medical history of their mothers regarding the use of various medications during pregnancy-such as estrogen, progesterone, thyroid hormones, antithyroid hormones, vitamins, microelements, and aspirin-will be examined. To facilitate this analysis, individual registration cards will be developed, approved by the ethics committee, and ratified by the Academic Council. The data will be submitted using Google Forms, followed by the inclusion of copyright information into the state register.
2. Evaluation of Anthropometric Data:

   This stage will assess the anthropometric data of 300 children under three years of age, focusing on those born after FET or fresh embryo transfer (Fresh-ET). Measurements will include weight, height, and head and chest circumference at the time of examination. Measurements for children under one year will utilize scales with a pan balance, a horizontal stadiometer, and a measuring tape. For children over one year, floor electronic scales, a vertical stadiometer, and a centimeter tape will be employed. Birth anthropometric data will be sourced retrospectively, while the WHO Child Growth Standards will be utilized to evaluate weight, height, head, and chest circumference relative to age and gender.
3. Study of Psychomotor Development:

   The psychomotor development of the 300 children under three years of age conceived via IVF or ICSI in fresh or frozen cycles will be assessed. This evaluation will employ standardized instruments such as the R. Griffiths Mental Development Scale and Denver Developmental Screening Tests. For children under one year, neurosonography will be conducted to assess brain structures, and retrospective results for children over one year of age will be extracted from medical records.

   The assessment aims to determine the functions of the nervous system utilizing the aforementioned standardized scales, focusing on various developmental parameters, including motor skills, social adaptation, communication abilities, and play skills. Scores will be compiled to ascertain overall developmental levels. The Denver II developmental screening test is specifically designed to assess children from birth to six years of age. It enhances diagnostic capabilities and evaluates several critical parameters, including: 1) personal and social characteristics, which examine the child's interactions with others and their ability to meet personal needs; 2) the development of gross and fine motor skills; 3) the development of both motor and sensory speech; and 4) an assessment of the child's behavior during the evaluation process.

   In cases where children are identified as being in the "risk group," a consultation with a neurologist is planned to establish examination protocols and identify the etiopathogenetic basis for potential developmental disorders. Standard methods of neurological examination will be utilized to assess the development of motor, sensory, cognitive, speech, emotional, communicative, and behavioral parameters in conjunction with anamnestic data and the overall state of somatic health.
4. Assessment of Reproductive Health:

The study will also evaluate the effect of ICSI, particularly in cases of male infertility, on the reproductive health and development of 200 male children under three years of age, in comparison with children conceived via classic IVF. This evaluation will involve objective examinations conducted by a pediatric andrologist to investigate the prevalence of urogenital pathology, supplemented by ultrasounds of the scrotum, kidneys, and bladder. Additionally, hormonal status will be assessed by Inhibin B and Anti-Müllerian Hormone (AMH). Anamnestic data will be collected to explore the relationship between the reproductive health of fathers and their sons born after ICSI.

3) Methods of Data Collection and Processing Data Collection Sources of Information: Data will be sourced from the International clinical center of the reproductology "PERSONA" and Institute of Reproductive Medicine (IRM clinic), in addition to direct examinations of participants based

DETAILED DESCRIPTION:
2.1. Introduction The forthcoming scientific and technical project aims to investigate the physical, cognitive, and reproductive health of children conceived by advanced ART methods. By examining this expanding cohort of children in Kazakhstan and conducting a comprehensive health assessment, the project seeks to elucidate the potential implications of advanced ART techniques on the incidence of future health issues in these offspring. The findings from this study will enable proactive identification and intervention for any potential health deviations, ensuring appropriate referrals to specialists for further evaluation and treatment.

2.2. The project objective: To enhance the management strategies for children conceived via ART, informed by the study of the impact of modern conception methods on the health of the offspring, and the formulation of management principles tailored to this population.

2.3. Project Tasks:

To attain the overall project goal, the following tasks must be addressed:

1. Analyze the influence of utilizing cryopreserved embryos in ART programs on the anthropometric characteristics and somatic health status of the offspring.
2. Investigate the neurological condition of children under three years of age conceived by advanced assisted reproductive techniques (ICSI and FET).
3. Evaluate the prevalence of urogenital pathology and hormonal profiles in male children under three years of age who were born using the ICSI method due to male factor infertility, in comparison to those conceived through classic IVF.
4. Examine the relationship between the reproductive health of fathers and their sons born after ICSI.
5. Assess the health status of children under three years of age born after successful ART programs, incorporating anamnestic data from their mothers, including medication usage before and during pregnancy.
6. Develop a predictive model and management algorithms for children conceived by various ART methods.

Rationale for Objectives:

1. Multidisciplinary Approach: The study integrates elements from reproductive science, gynecology, neonatology, andrology, urology, and pediatrics to understand ART's impact on offspring health comprehensively.
2. Focus on Advanced ART Methods: Emphasis will be placed on the outcomes associated with advanced assisted reproductive techniques, representing a significant contribution to the existing body of knowledge.
3. Comprehensive Health Assessment: The study will investigate diverse health metrics, including anthropometric characteristics, psychomotor development, and reproductive health of children conceived via advanced ART methods.
4. Geographical Considerations: This investigation stands as the first to analyze children conceived by advanced assisted reproductive techniques within Kazakhstan, considering unique socio-demographic factors.
5. Clinical Practice Improvement:: An in-depth examination of the characteristics of this demographic and identification of risk factors associated with pathological conditions will serve as valuable tools for enhancing outcomes in children conceived with advanced ART methods. The insights garnered from this study will contribute to improved counseling quality and a reduction in the financial burden associated with managing potential health complications in this population.

Following the completion of the project and the fulfillment of all designated tasks, the technological readiness level is anticipated to be 2. It will be attributed to the project's scientific and technical outcomes, which include the creation of a predictive model and the establishment of general principles for the care and management of children conceived by IVF or ICSI, utilizing either fresh or frozen cycles. Additionally, the project aims to publish articles based on the findings of applied research in peer-reviewed scientific journals that are indexed by international citation systems.

3. Scientific Novelty and Significance of the Project

1. Prerequisites for Project Development. The scientific novelty and significance of this project stem from the increasing acceptance and utilization of IVF as a viable method for addressing infertility. The enhanced accessibility and success rates of IVF procedures, coupled with socio-demographic trends such as delayed parenthood, have resulted in a substantial rise in the number of children born after ART. The provision of reimbursed 7,000 IVF cycles annually in Kazakhstan highlights the government's considerable focus on addressing infertility issues. Nevertheless, despite advancements in ART, the implications of advanced reproductive techniques on the health of offspring remain inadequately explored. Over recent decades, ART has experienced considerable evolution, paralleling developments in reproductive medicine. The adoption of FET and ICSI techniques has escalated significantly, raising concerns regarding their potential impact on offspring health. Research indicates that FET may contribute to the birth of large-for-gestational-age children and is associated with heightened risks of adverse obstetric and perinatal outcomes, as well as respiratory, infectious, and neurological disorders.

   Given the critical role of the sperm epigenome during early embryogenesis, it is imperative to scrutinize the consequences of utilizing sperm from men with infertility in ICSI procedures. Consequently, there is an increasing focus on the health status, endocrine, and reproductive profiles of boys and young adult males who were conceived by ICSI. While the literature has extensively documented the growth and overall health of children treated with ICSI, there is limited information regarding the gonadal function of these male offspring. Reports indicate occurrences of elevated genital malformations, diminished testosterone levels, and abnormal levels of Inhibin B and follicle-stimulating hormone (FSH) in boys conceived through ICSI. Inhibin B is pivotal in regulating the hypothalamic-pituitary-gonadal hormonal axis during childhood and measuring its serum levels in boys may provide significant clinical insights into potential deficiencies in gonadal development that may not manifest until puberty or later stages of life.

   Numerous studies underscore the potential association between prolonged use of high doses of hormonal medications in IVF programs and the emergence of metabolic disorders in offspring, including insulin resistance and prediabetes. Furthermore, there is an increased risk of inflammatory conditions in children, which may present as a higher incidence of infectious diseases during early childhood. An additional critical consideration is the impact of medications administered for concomitant conditions in women undergoing IVF. For instance, the use of antithyroid medications during early pregnancy has been consistently linked to an elevated risk of congenital anomalies. The mechanisms underlying the teratogenic effects of these agents require further investigation, although they are presumably related to disruptions in thyroid hormonal regulation during pivotal stages of embryogenesis. Concerns have also been raised regarding the potential increase in the risk of malformations associated with dydrogesterone in the first trimester of pregnancy; however, further research is necessary to substantiate this correlation and elucidate the dose-dependent nature of the effect.

   The influence of ART on the neurodevelopmental outcomes of offspring warrants particular attention. The current literature reveals a dearth of specific studies assessing long-term cognitive, behavioral, and mental health effects in children conceived by ART, thus limiting our comprehension of possible repercussions. Moreover, there is a notable prevalence of perinatal complications in children born after ART, including hypoxic-ischemic brain injury and pathological hyperbilirubinemia, which may significantly affect the child's future health and development.
2. Justification of Scientific Novelty Existing data are limited but suggest that modern techniques, paternal infertility, and maternal pharmacological interventions during gestation may contribute to certain adverse health outcomes in offspring. The objective of our project is to address these gaps by conducting a study that encompasses innovative assisted reproductive techniques and assesses not only the physical and neuropsychiatric outcomes but also the reproductive health of children born after ART in Kazakhstan. The findings from this investigation will enhance understanding of the implications of utilizing advanced techniques, thereby facilitating improvements in ART guidelines, clinical practices, and the mitigation of potential risks to offspring, as well as the development of management algorithms. The proposed study of a cohort of children in Kazakhstan has the potential to significantly augment the existing database and enhance the reliability of the findings, allowing for more generalized conclusions that may be applicable at a global level.

The novelty of this study lies in its comprehensive analysis of the effects of advanced ART methods, including ICSI and FET on the health status and development of offspring. By examining the somatic, neuropsychological, and reproductive health of children conceived by these methods, the research offers new insights into the potential risks and outcomes linked to ART.

4) Impact of the Project This project, which is dedicated to the long-term examination of the implications of advanced ART methods on offspring health, holds significant socio-economic relevance for Kazakhstan. Its scope transcends mere medical inquiry, addressing fundamental aspects of national well-being. The recommendations developed through this project for optimizing ART guidelines and implementing postnatal monitoring for children conceived via advanced technologies will have practical applications within Kazakhstan's healthcare framework. This initiative will facilitate the timely identification and effective treatment of potential pathological conditions, thereby reducing morbidity and mortality rates among children conceived by ART.

Furthermore, the emphasis on early diagnosis and preventative measures has the potential to substantially lower the costs associated with long-term treatment and rehabilitation. The anticipated economic benefits will also alleviate pressure on the healthcare system. The importance of this project extends beyond the medical realm; it exemplifies Kazakhstan's commitment to investing in scientific research and advancing healthcare development, which is essential for enhancing the quality of life for its population and bolstering the country's reputation on the global stage.

The findings of this study will be disseminated widely among the medical community and the public, thereby enhancing awareness of ART and improving the reproductive health landscape. The successful completion of this project will serve as a model for other nations seeking to refine their reproductive health systems and elevate the standard of healthcare for all citizens. Additionally, the data generated may be instrumental in formulating national programs dedicated to reproductive health and offering support for families with children conceived by ART. Ultimately, this initiative contributes to the social well-being and economic development of Kazakhstan, ensuring a healthy future for subsequent generations.

4. Research Methods and Ethical Issues

1. Main Scientific Questions and Hypotheses of the Project The primary objective of this project is to investigate the impact of advanced ART methods on the health status of children. The central scientific questions being addressed include: What are the consequences of ICSI and FET on the physical, cognitive, and reproductive health of children? The underlying hypothesis posits that children conceived by advanced ART methods may present with health indicators that deviate from the established norms.
2. Description of the Experiments

Research Methods:

To achieve the goals of the study, the following stages are anticipated:

1. Retrospective Analysis of Anamnestic Data:

   This stage involves studying the relationship between the physical status and morbidity structure of 300 children under the age of three, who were conceived by advanced ART methods. Additionally, the medical history of their mothers regarding the use of various medications during pregnancy-such as estrogen, progesterone, thyroid hormones, antithyroid hormones, vitamins, microelements, and aspirin-will be examined. To facilitate this analysis, individual registration cards will be developed, approved by the ethics committee, and ratified by the Academic Council. The data will be submitted using Google Forms, followed by the inclusion of copyright information into the state register.
2. Evaluation of Anthropometric Data:

   This stage will assess the anthropometric data of 300 children under three years of age, focusing on those born after FET or fresh embryo transfer (Fresh-ET). Measurements will include weight, height, and head and chest circumference at the time of examination. Measurements for children under one year will utilize scales with a pan balance, a horizontal stadiometer, and a measuring tape. For children over one year, floor electronic scales, a vertical stadiometer, and a centimeter tape will be employed. Birth anthropometric data will be sourced retrospectively, while the WHO Child Growth Standards will be utilized to evaluate weight, height, head, and chest circumference relative to age and gender.
3. Study of Psychomotor Development:

   The psychomotor development of the 300 children under three years of age conceived via IVF or ICSI in fresh or frozen cycles will be assessed. This evaluation will employ standardized instruments such as the R. Griffiths Mental Development Scale and Denver Developmental Screening Tests. For children under one year, neurosonography will be conducted to assess brain structures, and retrospective results for children over one year of age will be extracted from medical records.

   The assessment aims to determine the functions of the nervous system utilizing the aforementioned standardized scales, focusing on various developmental parameters, including motor skills, social adaptation, communication abilities, and play skills. Scores will be compiled to ascertain overall developmental levels. The Denver II developmental screening test is specifically designed to assess children from birth to six years of age. It enhances diagnostic capabilities and evaluates several critical parameters, including: 1) personal and social characteristics, which examine the child's interactions with others and their ability to meet personal needs; 2) the development of gross and fine motor skills; 3) the development of both motor and sensory speech; and 4) an assessment of the child's behavior during the evaluation process.

   In cases where children are identified as being in the "risk group," a consultation with a neurologist is planned to establish examination protocols and identify the etiopathogenetic basis for potential developmental disorders. Standard methods of neurological examination will be utilized to assess the development of motor, sensory, cognitive, speech, emotional, communicative, and behavioral parameters in conjunction with anamnestic data and the overall state of somatic health.
4. Assessment of Reproductive Health:

The study will also evaluate the effect of ICSI, particularly in cases of male infertility, on the reproductive health and development of 200 male children under three years of age, in comparison with children conceived via classic IVF. This evaluation will involve objective examinations conducted by a pediatric andrologist to investigate the prevalence of urogenital pathology, supplemented by ultrasounds of the scrotum, kidneys, and bladder. Additionally, hormonal status will be assessed by Inhibin B and Anti-Müllerian Hormone (AMH). Anamnestic data will be collected to explore the relationship between the reproductive health of fathers and their sons born after ICSI.

3) Methods of Data Collection and Processing Data Collection Sources of Information: Data will be sourced from the International clinical center of the reproductology "PERSONA" and Institute of Reproductive Medicine (IRM clinic), in addition to direct examinations of participants based on the Persona Clinic framework. This strategy is designed to ensure the acquisition of comprehensive and accurate information regarding the health of children, in conjunction with their parents' medical histories.

Methods of Data Collection: The data collection process will encompass history taking, conducting clinical examinations, and performing laboratory and instrumental studies. The inclusion criteria will involve subjects who have successfully undergone ART programs after IVF and ICSI, specifically involving the transfer of fresh or cryopreserved embryos. Exclusion criteria will encompass intrauterine insemination utilizing sperm from either the female participant's partner or a sperm donor, as well as programs employing donor gametes and surrogacy arrangements.

Data Processing The statistical analysis of the collected data will be executed using Microsoft Excel 2016 and the advanced statistical methodology provided by IBM SPSS Statistics 26. Both parametric and nonparametric statistical techniques will be employed. Descriptive statistics will involve the calculation of the arithmetic mean and standard error of the mean. The comparison of mean values between two independent groups will be facilitated through the Mann-Whitney U test (for nonparametric data) or the Student's t-test (for parametric data). Frequency data analysis, such as the examination of disease incidence in children relative to risk factors, will be conducted utilizing the Pearson χ² test or Fisher's exact test. Additionally, binary logistic regression will serve to analyze the influence of multiple independent variables on a binary outcome (e.g., presence or absence of a disease). The efficacy of the logistic regression model will be evaluated through ROC analysis to ascertain the optimal cutoff threshold and to assess the diagnostic value of the model. The sensitivity and specificity of the diagnostic test will be computed to evaluate its diagnostic accuracy. Results will be systematically presented in tables and graphs, accompanied by a detailed narrative in the study report. The findings of the study will be rooted in statistically significant results and contextualized within the existing literature. The data generated will facilitate the formulation of recommendations aimed at the prevention and early detection of diseases in children associated with prenatal factors. Differences observed between the compared groups will be regarded as statistically significant at a p-value threshold of less than 0.05.

4) Principles and Norms of Scientific Ethics This project places significant emphasis on ethical considerations, particularly regarding the handling of confidential data concerning children. We acknowledge the heightened responsibility associated with research that impacts the health of minors and adhere rigorously to the highest ethical standards recognized in international practice. This adherence includes obtaining mandatory informed consent from parents or legal guardians for the participation of their children in the study, as well as ensuring the protection of personal data. All collected information will be anonymized and stored on secure servers with restricted access, thereby mitigating the risk of unauthorized access or disclosure. The research methodology will undergo thorough review to ensure compliance with the principles of fairness, beneficence, and respect for the individual, thereby safeguarding the rights and welfare of both the children involved and their families. Scientific integrity will be a cornerstone of our research, and all findings will be meticulously verified for accuracy and reliability prior to publication. The procedures and methodologies employed in the planned studies will fully adhere to the legislation of the Republic of Kazakhstan.

ELIGIBILITY:
Inclusion Criteria:

For children:

* Born as a result of an ART program (IVF, ICSI, FET, or Fresh-ET).
* Age at the time of assessment: from birth up to 36 months.
* Availability of complete perinatal and medical documentation, including ART cycle characteristics and neonatal outcomes.
* Informed consent provided by parents or legal guardians for participation in the study and for biological sample collection (where applicable).

For mothers:

* History of pregnancy achieved through ART within the territory of Kazakhstan.
* Availability of data on pharmacological treatment before and during pregnancy (e.g., hormonal therapy, antithyroid drugs, vitamins, micronutrients).
* Willingness to provide anamnestic and perinatal information, and consent for access to medical records.

For fathers (in ICSI subgroup):

* Documented infertility factor necessitating ICSI.
* Agreement to provide relevant medical history and participate in comparative analyses (e.g., endocrine or reproductive parameters of father-son pairs).

Ages: 0 Months to 3 Years | Sex: All
Age Groups: Child
Study Population: The study population will consist of children under three years of age who were conceived via assisted reproductive technologies (ART) in the Republic of Kazakhstan, along with their biological parents.
  The research cohort will include children conceived through advanced ART methods - specifically intracytoplasmic sperm injection (ICSI) and frozen embryo transfer (FET) - as well as a comparison group of children conceived via conventional IVF and fresh embryo transfer (Fresh-ET).
  A total of approximately 300 children (including at least 200 male participants for reproductive health analysis) will be recruited from reproductive medicine centers, pediatric hospitals, and outpatient clinics across Kazakhstan. Medical records of participating mothers will also be used for retrospective data collection regarding conception details, pregnancy course, and perinatal outcomes.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Physical growth parameters of children conceived via ART (ICSI and FET) | At birth (medical records) and at clinical assessment conducted at the child's age at enrollment (up to 36 months of age).
  Evaluation of physical growth using standardized anthropometric measures: weight (kg), length/height (cm), and head circumference (cm), assessed against WHO Child Growth Standards.
  Unit of Measure:
  Z-scores (weight-for-age, length-for-age, head-circumference-for-age).
Psychomotor and neurodevelopmental status of children conceived via ART (ICSI and FET) | At a single clinical assessment conducted at the child's age at enrollment (up to 36 months of age).
  Assessment of cognitive, motor, language, and social-emotional development using the Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-IV).
  Scores range from 40 to 160; higher scores indicate better developmental performance.
  Unit of Measure:
  Bayley-IV composite scores (Cognitive, Motor, Language).
Urogenital and reproductive system development in children conceived via ART (ICSI and FET) | At a single clinical assessment conducted at the child's age at enrollment (up to 36 months of age).
  Clinical examination and ultrasonographic assessment of urogenital system development performed by pediatric urologists/gynecologists.
  Parameters include presence or absence of congenital anomalies (e.g., cryptorchidism, hypospadias), uterus/ovary/testis morphology, and developmental measurements as per pediatric normative standards.
  Unit of Measure:
  Incidence of anomalies (yes/no), organ measurements (mm).

SECONDARY OUTCOMES:
Weight-for-Age Z-Score | At birth (medical records) and at clinical assessment conducted at the child's age at enrollment (up to 36 months of age).
  Assessment of somatic growth using WHO Child Growth Standards.
Height-for-Age Z-Score | At birth (medical records) and at clinical assessment conducted at the child's age at enrollment (up to 36 months of age).
  Evaluation of linear growth relative to age-specific WHO standards.
Head Circumference-for-Age Z-Score | At birth (medical records) and at clinical assessment conducted at the child's age at enrollment (up to 36 months of age).
  Measurement of head growth relative to WHO Child Growth Standards.
Psychomotor development score (Griffiths Scales) | At a single clinical assessment conducted at the child's age at enrollment (up to 36 months of age).
  Global developmental assessment using the Griffiths Mental Development Scales, including motor, communication, social, and cognitive domains.
  Assessment Tool: Griffiths Mental Development Scales (GMDS). Range: Developmental Quotient (DQ), typically 0-130; higher scores indicate better developmental performance.
  Unit of Measure: Griffiths DQ Composite Score.
Developmental screening result (Denver II Test) | At a single clinical assessment conducted at the child's age at enrollment (up to 36 months of age).
  Screening for developmental delays in four domains (personal-social, fine motor-adaptive, language, gross motor).
  Assessment Tool: Denver II Developmental Screening Test. Outcome Categories: Pass / Fail / Caution. Unit of Measure: Denver II Classification.
Presence of neurosonography abnormalities | At a single assessment conducted at the child's age at enrollment (up to 12 months), or extracted from existing medical records if the examination was previously performed.
  Identification of abnormalities in brain structures among children <12 months.
Prevalence of urogenital abnormalities | At a single clinical assessment conducted at the child's age at enrollment (up to 36 months of age).
  Evaluation of structural findings on pediatric andrological examination and ultrasound (scrotum, kidneys, bladder).
Serum Inhibin B concentration | At a single clinical assessment conducted at the child's age at enrollment (up to 36 months of age).
  Evaluation of early reproductive function in male children conceived via different ART methods.
  Unit of Measure: pg/mL.
Serum AMH (Anti-Müllerian Hormone) concentration | At a single clinical assessment conducted at the child's age at enrollment (up to 36 months of age).
  Assessment of Sertoli cell function in male children. Unit of Measure: pg/mL.
Association between parental medical history and offspring health parameters | At the child's enrollment visit (up to 36 months of age), using parental medical history collected at the same visit or extracted from medical records.
  Exploratory analysis of maternal medication use and paternal reproductive factors in relation to child growth, neurodevelopment, and reproductive outcomes.
  Unit of Measure: Statistical association (multivariate model coefficients; no direct clinical measurement).

CONTACTS AND LOCATIONS:
Locations (1):
- Международный клинический центр репродуктологии Persona, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: No
Because the study involves minors, sensitive reproductive and health data, and national medical records, sharing individual participant data (IPD) outside the research institution would raise ethical and privacy concerns. Additionally, Kazakhstan's current biomedical research regulations typically restrict data transfer abroad or to third parties without explicit consent and data-sharing agreements.